CLINICAL TRIAL: NCT07023627
Title: A Phase 2, Single-Arm Study of INCB123667 in Participants With Platinum-Resistant Ovarian Cancer With Cyclin E1 Overexpression (MAESTRA 1)
Brief Title: A Study of INCB123667 in Participants With Platinum-Resistant Ovarian Cancer With Cyclin E1 Overexpression
Acronym: MAESTRA 1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Collaborators: ENGOT Foundation (Unknown); GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB123667-203; GOG-3129 (Other: GOG Study Number); 2025-521513-14-00 (Registry Identifier: EU CT Number); OV94 (Other: ENGOT Study Number)
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Ovarian Cancer
Keywords: INCB123667
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): INCB123667 will be administered at the protocol defined dose based on their tumor cyclin E1 expression levels as defined in the protocol.
  Interventions: Drug: INCB123667
- Cohort 2 (Experimental): INCB123667 will be administered at the protocol defined dose based on their tumor cyclin E1 expression levels as defined in the protocol.
  Interventions: Drug: INCB123667
- Cohort 3 (Experimental): INCB123667 will be administered at the protocol defined dose based on their tumor cyclin E1 expression levels as defined in the protocol.
  Interventions: Drug: INCB123667

INTERVENTIONS:
Drug: INCB123667 — Administered orally twice daily (BID).

SUMMARY:
This study will evaluate the safety and efficacy of INCB123667 in Participants With Platinum-Resistant Ovarian Cancer (PROC) With Cyclin E1 Overexpression.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of a high-grade serous epithelial ovarian, fallopian tube, or primary peritoneal cancer.
* Have platinum-resistant disease:

  * Participants who have only had 1 line of platinum-based therapy must have received at least 4 cycles of a platinum-containing regimen.
  * Participants who have received 2 to 4 lines of platinum-based therapy must have progressed on or within 6 months after the last dose of platinum.
* Willingness to undergo a pretreatment biopsy. Note: Tissue from a fresh pretreatment biopsy is preferred, however an archival sample is acceptable as long as the sample is no older than 5 years.
* Received at least 1 and no more than 4 prior lines of systemic therapy following the initial diagnosis, after which single-agent therapy is considered an appropriate next therapeutic option.
* Must have received bevacizumab unless there was a contraindication for its use.
* If the tumor tests positive for FRα, participants must have received mirvetuximab soravtansine unless there is an exception for its use on medical grounds.

Exclusion Criteria:

* Have endometrioid, clear cell, mucinous, or sarcomatous histology, mixed tumors containing any of these histologies, or low-grade/borderline ovarian cancer.
* Have primary platinum-refractory disease: either did not respond (CR or PR) to first-line platinum-containing therapy or progressed on or within 3 months after the last dose of the first line platinum-containing therapy.
* The tumor tests positive for FRα but the participant has not received mirvetuximab soravtansine for any reason other than medical contraindication.
* Clinically significant or uncontrolled cardiac disease within 6 months before the first dose of study drug.
* Known active CNS metastases and/or carcinomatous meningitis.
* Known additional malignancy that is progressing or requires active treatment.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2027-04-27 (Estimated); Study Completion 2027-10-24 (Estimated)

PRIMARY OUTCOMES:
Objective Response by IRC | Up to 2 years
  Defined as having a confirmed best overall response of complete response (CR) or partial response (PR), as determined by independent review committee (IRC) assessment per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Duration of Response (DOR) by IRC | Up to 2 years
  Defined as the time from the earliest date of CR or PR contributing to a subsequently confirmed CR or PR until the earliest date of disease progression, as determined by IRC assessment per RECIST v1.1, or death due to any cause, whichever occurs first.
Progression-Free Survival (PFS) by IRC | Up to 2 years
  Defined as the time from the date of first dose of study drug until the earliest date of disease progression as determined by IRC assessment per RECIST v1.1, or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to 2 years
  Defined as the time from the date of first dose of study drug until death due to any cause.
Objective Response by Investigator | Up to 2 years
  Defined as having a confirmed best overall response of CR or PR, as determined by investigator assessment per RECIST v1.1.
DOR by investigator | Up to 2 years
  Defined as the time from the earliest date of CR or PR contributing to a subsequently confirmed CR or PR until the earliest date of disease progression, as determined by investigator assessment per RECIST v1.1, or death due to any cause, whichever occurs first.
PFS by Investigator | Up to 2 years
  Defined as the time from the date of first dose of study drug until the earliest date of disease progression, as determined by investigator assessment per RECIST v1.1, or death due to any cause, whichever occurs first.
Treatment Emergent Adverse Events (TEAE'S) | Up to 2 years and 30 days
  Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug until 30 days after the last dose of study drug or the start of new anticancer therapy, whichever occurs first.
TEAEs leading to dose interruptions, dose reductions or discontinuation of study treatment | Up to 2 years and 30 days
  TEAEs leading to dose interruptions, dose reductions or discontinuation of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (80):
- United States (41):
  - Usa Health Mitchell Cancer Institute, Mobile, Alabama
  - Uams Winthrop P Rockefeller Cancer Institute, Little Rock, Arkansas
  - University of California, Los Angeles Medical Center, Los Angeles, California
  - Scripps Healthscripps Mercy Hospital Prebys Cancer Center, San Diego, California
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Florida Cancer Specialists & Research Institute, Fort Myers, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Florida Cancer Specialists & Research Institute, West Palm Beach, Florida
  - Northeast Georgia Medical Center Gainesville, Gainesville, Georgia
  - Parkview Research Center, Fort Wayne, Indiana
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Norton Cancer Institute, Louisville, Kentucky
  - Trials365, Llc, Shreveport, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - John Hopkins University-School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Umass Memorial Medical Center, Inc., Worcester, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Minnesota Oncology-Minneapolis, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University, St Louis, Missouri
  - St. Vincent Regional Hospital - West End Clinic, Billings, Montana
  - Methodist Hospital Methodist Estabrook Cancer Center, Omaha, Nebraska
  - John Theurer Cancer Center, Hackensack University Medical Center, Hackensack, New Jersey
  - Laura and Isaac Perlmutter Cancer Center, New York, New York
  - State University of New York Upstate Medical Unive, Syracuse, New York
  - Oncology Hematology Care, Inc, Cincinnati, Ohio
  - The Mark H Zangmeister Cancer Center Ohio, Columbus, Ohio
  - The Ohio State University Wexner Medical Center Division of Gynecologic Oncology, Hilliard, Ohio
  - Penn State College of Medicine, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Oncology-Austin Center, Austin, Texas
  - Cancer Care Center of South Texas-Medical Center, San Antonio, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Virginia Cancer Specialists, Pc, Fairfax, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - West Virginia University, Morgantown, West Virginia
  - Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (6):
  - Blacktown Cancer & Haematology Centre-Blacktown Hospital, Blacktown, New South Wales
  - Concord General Repatriation Hospital, Concord, New South Wales
  - Burnside War Memorial Hospital - the Brian Fricker Oncology Centre, Adelaide, South Australia
  - Hobart Hospital-Royal Hobart Hospital, Hobart, Tasmania
  - Cancer Research Sa (Crsa), Adelaide
  - Southern Oncology Clinical Research Unit, South Australia
- Belgium (5):
  - Hopital Universitaire de Bruxelles (Academisch Ziekenhuis Brussel), Brussels
  - Cliniques Universitaires St Luc Ucl, Brussels
  - Az Groeninge Campus Kennedylaan, Kortrijk
  - Universitair Ziekenhuis Leuven, Leuven
  - Chu Liege, Liège
- Japan (7):
  - Hyogo Cancer Center, Akashi-shi
  - Saitama Medical University International Medical Center, Hidaka-shi
  - The Cancer Institute Hospital of Jfcr, Kōtoku
  - Kurume University Hospital, Kurume
  - Nho Shikoku Cancer Center, Matsuyama
  - Hokkaido University Hospital, Sapporo Hokkaido
  - Shizuoka Cancer Center, Sunto-gun
- Panoncology Trials, San Juan, PR, Puerto Rico
- Spain (10):
  - Hospital Universitario Vall D'Hebron, Barcelona
  - Hospital Clinic de Barcelona (Hospital Clinic I Provincial), Barcelona
  - Instituto Catalan de Oncologia - Hospital Duran I Reynals, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Institut Catala D'Oncologia Girona, Girona
  - Clinica Universidad de Navarra - Sede Madrid, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de La Arrixaca, Murcia
  - Instituto Valenciano de Oncologia, Valencia
  - Hospital Clinico Universitario de Valencia (Instituto de Investigacion Sanitaria Incliva), Valencia
- Switzerland (5):
  - Istituto Oncologico Della Svizzera Italiana, Bellinzona
  - Kantonsspital Graubunden, Chur
  - Geneva University Hospitals-Hug, Geneva
  - Centre Hospitalier Universitaire Vaudois Lausanne (Chuv) - Centre Du Cancer Lausanne-Batiment Hospit, Lausanne
  - Kantonsspital Baselland (Ksbl) - Standort Liestal - Medizinische Universitatsklinik, Liestal
- United Kingdom (5):
  - St Bartholomew'S Hospital, London
  - Guy'S Hospital - Guy'S & St Thomas' Nhs Foundation Trust, London
  - Royal Marsden Hospital (Sutton) - Royal Marsden Nhs Foundation Trust, London
  - Hammersmith Hospital - Imperial College Healthcare Nhs Trust, London
  - The Christie Nhs Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A study of INCB123667 in Participants With Platinum-Resistant Ovarian Cancer With Cyclin E1 Overexpression — https://incyteclinicaltrials.com/studies/incb123667-203